CLINICAL TRIAL: NCT05681208
Title: The Effect of Motivational Interview, Prepared According to the Health Behavior Interaction Model, on Microbiota Awareness and Attitudes on Infant Nutrition in Primiparous Mothers Who Start Complementary Nutrition: A Randomized Controlled Study
Brief Title: Microbiota Awareness and Nutrition Education Given to Mothers With Motivational Interview
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeşim Ceylantekin, Asst. Prof., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AfyonkarahisarHSU-YC-1
Record Dates: First submitted 2022-12-15; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Microbiota
Keywords: microbiota; motivational interview; health behavior interaction model
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The training, which is prepared based on the motivational interview method, will be given individually, starting when baby is 4 months old, will be interviewed once a week for nine weeks. In first meeting; before starting motivational interview, mothers were interviewed face-to-face with the Baby, Mother Introductory Information Form, Mothers', Babies' Food Consumption Frequency Registration Form, Microbiota Awareness Scale (MFI), Infant Nutrition Attitude Scale (LOWA), Behavior Change Stage Diagnostic Form, Motivational Interview rating the schedule will be applied. At the end of this meeting, which lasts for 45-50 minutes, next meeting date will be determined, the meeting will be terminated. Second interview is planned to last 60-90 minutes. After the second meeting, Motivational interviews will provide information on nutritional posters, brochures of the Ministry of Health, complementary nutrition, nutrition for microbiota. The scales to be used will be re-administered.
  Interventions: Behavioral: Motivational interview
- Control group (No Intervention): Within the scope of the research, no intervention will be made to the mothers in the control group other than routine family health center practices. In Turkey, 4-month-old baby follow-up continues at the Family Health Center, followed by midwives, nurses and doctors. Scales will be applied to mothers by face-to-face interview method when they come for routine baby follow-up. The training content given in the Family Health Center will be presented to the control group.

INTERVENTIONS:
Behavioral: Motivational interview — Information will be given about the motivational interviews to be held and the objectives and content of the motivational interviews will be explained clearly. Care will be taken to ensure that the content of the brochures and materials provided is not too dense. It was prepared according to the Health Behavior Interaction Model of motivational interview steps. The first meeting of the motivational interview will start in the 4th month and the meetings will continue to be held every week for the first month and a half, and every two weeks for the next month and a half.
  Negotiations will end in nine weeks. After the last interview, the scales will be applied to the mother again. Motivational interviews are planned to last 60-90 minutes (first session 45-50 minutes) every week.
  Arms: Intervention group

SUMMARY:
Complementary nutrition is considered a critical step not only for changes in nutritional requirements but also for the formation of life-long taste preferences, nutrition and eating habits that may affect health in the long run. While the microbiota is developing, in the early stages of life, the wrong food choice negatively affects the microbiota development and causes malnutrition. In this study, the effect of motivational interviews prepared according to the Health Behavior Interaction Model on microbiota awareness and infant feeding attitude will be investigated in primiparous mothers who will start complementary feeding.

ELIGIBILITY:
Inclusion Criteria:

* Mothers over the age of 18,
* Ability to read and write Turkish,
* Absence of any disease in the mother and child,
* The mother's willingness to participate in the research,
* Having a healthy, vaginal and mature delivery,
* Being a primiparous mother
* Feeding only with breast milk,

Exclusion Criteria:

Mothers not participating in at least one training,

* Mothers not participating in the motivational interview,
* Desire to leave the research
* Absence of ambivalent feelings
* Inability to create a food consumption frequency scheme

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers over 18
Enrollment: 64 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Microbiota awareness scale | before the 1st interview
  -Microbiota awareness scale total score (The score range of the scale was defined as the lowest 18 points and the highest 100 points. The cut-off score was not specified in the scale. The high score obtained from the scale was evaluated as a high level of microbiota awareness. The draft form of the scale was developed as a five-point Likert type (1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree) and includes 27 positive and 2 negative statements. Two of the questions in the scale are knowledge questions with five options, marking the correct one was evaluated as 1 point and not marking the wrong one was evaluated as 1 point. The last two questions consist of open-ended questions. Those who do not answer these questions are given 1 point, one answer is 2 points, two answers are 3 points, three answers are 4 points, and those who answer four or more are 5 points.
Microbiota awareness scale | Last follow-up after 5th interview (1 month after first meeting)
  * Microbiota awareness scale total score (The score range of the scale was defined as the lowest 18 points and the highest 100 points. The cut-off score was not specified in the scale. The high score obtained from the scale was evaluated as a high level of microbiota awareness.)
  * General information sub-dimension score level
  * Product information sub-dimension score level
  * Chronic disease sub-dimension score level
  * Probiotic and prebiotic sub-dimension score level
Microbiota awareness scale | Last follow-up after 9th interview(1 month after the second interview)
  * Microbiota awareness scale total score (The score range of the scale was defined as the lowest 18 points and the highest 100 points. The cut-off score was not specified in the scale. The high score obtained from the scale was evaluated as a high level of microbiota awareness).
  * General information sub-dimension score level
  * Product information sub-dimension score level
  * Chronic disease sub-dimension score level
  * Probiotic and prebiotic sub-dimension score level